CLINICAL TRIAL: NCT00041444
Title: Multi-Ethnic Study of Atherosclerosis-Eye Study
Brief Title: Multi-Ethnic Study of Atherosclerosis (MESA) - Ancillary Eye Study
Acronym: MESA-Eye
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2001-409; R01HL069979 (NIH); 1182 (Other: Study Team)
Record Dates: First submitted 2002-07-08; First posted 2002-07-09 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Coronary Arteriosclerosis; Coronary Disease; Cerebrovascular Disorders; Heart Failure, Congestive; Myocardial Infarction; Heart Diseases; Diabetes Mellitus, Non-insulin Dependent; Hypertension; Diabetic Retinopathy; Macular Degeneration; Diabetes Mellitus
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease; Cerebrovascular Disorders; Heart Failure; Myocardial Infarction; Heart Diseases; Diabetes Mellitus, Type 2; Hypertension; Diabetic Retinopathy; Macular Degeneration; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To evaluate the relation of retinal microvascular characteristics to subclinical cardiovascular disease, clinical disease, and their risk factors in the Multi-Ethnic Study of Atherosclerosis (MESA) cohort.

DETAILED DESCRIPTION:
BACKGROUND:

The study further expands and enlarges the findings of the NHLBI-supported Atherosclerosis Risk in Communities (ARIC) study on the relationship of retinal microvascular disease to the presence of subclinical and clinical cardiovascular disease among Multi-Ethnic Study of Atherosclerosis (MESA) participants. ARIC data showed that retinal microvascular changes were associated with the following findings: markers of persistent hypertensive damage, markers of inflammation and endothelial dysfunction, magnetic resonance imaging (MRI)-detected cerebral infarct independent of hypertension, predictive of 3-year incident stroke independent of hypertension, and predictive of 3-year incident coronary heart disease in women but not men.

DESIGN NARRATIVE:

The MESA-EYE study is a separate add-on to the Multi-Ethnic Study of Atherosclerosis, a six regional center 10 year program begun in July 2000. The overall goals of the parent study are the identification of risk factors for subclinical cardiovascular disease, for progression of subclinical disease, and for transition of subclinical to clinical cardiovascular disease. The eye component will tie in with Exam 2 of the main study which begins August 2002 and runs through January 2004. Retinal photography to document microvascular changes will be performed on the approximately 6,500 MESA participants at Exam 2. Retinal photography will follow a standardized written protocol similar to that used in ARIC. Focal arterial narrowing and AV nicking will be classified as definite, questionable, or none. Data handling will be based on protocols previously used in several other NIH sponsored clinical trials where eye retinal studies were performed.

The six specific aims of the study are to: (1) determine the relationship of retinal microvascular characteristics to measures of subclinical CVD through (a) magnetic resonance imaging of left ventricular function (b) brachial artery ultrasound for flow mediated endothelial vasodilatation (c) radial artery tonometry measurement of peripheral artery function (d) magnetic resonance imaging for myocardial perfusion; (2) determine relationship of retinal microvascular characteristics to clinical CVD, specifically: (a) coronary heart disease (b) congestive cardiac failure (c) stroke; (3) determine relationship of retinal microvascular characteristics to CVD risk factors, specifically:(a) development of type 2 diabetes (b) development of hypertension (c) markers of: (I) inflammation (II) hemostasis (III) fibrinolysis; (4) determine the relation of retinal microvascular changes to structural and functional disorders of the brain; (5) describe the prevalence of retinal microvascular abnormalities in different racial/ethnic groups; (6) describe the prevalence and risk factors of (a) diabetic retinopathy (b) age-related maculopathy.

ELIGIBILITY:
No eligibility criteria

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6176 (Actual)
Dates: Start 2002-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Klein, MD, MPH, Principal Investigator — University of Wisconsin, Madison

REFERENCES:
- [Result] Klein R, Meuer SM, Moss SE, Klein BE, Neider MW, Reinke J. Detection of age-related macular degeneration using a nonmydriatic digital camera and a standard film fundus camera. Arch Ophthalmol. 2004 Nov;122(11):1642-6. doi: 10.1001/archopht.122.11.1642. PMID 15534124
- [Result] Fernandez AB, Wong TY, Klein R, Collins D, Burke G, Cotch MF, Klein B, Sadeghi MM, Chen J. Age-related macular degeneration and incident cardiovascular disease: the Multi-Ethnic Study of Atherosclerosis. Ophthalmology. 2012 Apr;119(4):765-70. doi: 10.1016/j.ophtha.2011.09.044. Epub 2011 Dec 23. PMID 22197438
- [Result] Adar SD, Klein R, Klein BE, Szpiro AA, Cotch MF, Wong TY, O'Neill MS, Shrager S, Barr RG, Siscovick DS, Daviglus ML, Sampson PD, Kaufman JD. Air Pollution and the microvasculature: a cross-sectional assessment of in vivo retinal images in the population-based multi-ethnic study of atherosclerosis (MESA). PLoS Med. 2010 Nov 30;7(11):e1000372. doi: 10.1371/journal.pmed.1000372. PMID 21152417
- [Result] Cheung N, Sharrett AR, Klein R, Criqui MH, Islam FM, Macura KJ, Cotch MF, Klein BE, Wong TY. Aortic distensibility and retinal arteriolar narrowing: the multi-ethnic study of atherosclerosis. Hypertension. 2007 Oct;50(4):617-22. doi: 10.1161/HYPERTENSIONAHA.107.091926. Epub 2007 Aug 13. PMID 17698721
- [Result] Cheung N, Islam FM, Jacobs DR Jr, Sharrett AR, Klein R, Polak JF, Cotch MF, Klein BE, Ouyang P, Wong TY. Arterial compliance and retinal vascular caliber in cerebrovascular disease. Ann Neurol. 2007 Dec;62(6):618-24. doi: 10.1002/ana.21236. PMID 17918248
- [Result] Klein R, Li X, Kuo JZ, Klein BE, Cotch MF, Wong TY, Taylor KD, Rotter JI. Associations of candidate genes to age-related macular degeneration among racial/ethnic groups in the multi-ethnic study of atherosclerosis. Am J Ophthalmol. 2013 Nov;156(5):1010-1020.e1. doi: 10.1016/j.ajo.2013.06.004. Epub 2013 Aug 12. PMID 23938121
- [Result] Wong TY, Klein R, Islam FM, Cotch MF, Folsom AR, Klein BE, Sharrett AR, Shea S. Diabetic retinopathy in a multi-ethnic cohort in the United States. Am J Ophthalmol. 2006 Mar;141(3):446-455. doi: 10.1016/j.ajo.2005.08.063. PMID 16490489
- [Result] Klein R, Knudtson MD, Klein BE, Wong TY, Cotch MF, Barr G. Emphysema, airflow limitation, and early age-related macular degeneration. Arch Ophthalmol. 2010 Apr;128(4):472-7. doi: 10.1001/archophthalmol.2010.25. PMID 20385944
- [Result] Colagiuri S, Lee CM, Wong TY, Balkau B, Shaw JE, Borch-Johnsen K; DETECT-2 Collaboration Writing Group. Glycemic thresholds for diabetes-specific retinopathy: implications for diagnostic criteria for diabetes. Diabetes Care. 2011 Jan;34(1):145-50. doi: 10.2337/dc10-1206. Epub 2010 Oct 26. PMID 20978099
- [Result] Klein R, Knudtson MD, Klein BE, Wong TY, Cotch MF, Liu K, Cheng CY, Burke GL, Saad MF, Jacobs DR Jr, Sharrett AR. Inflammation, complement factor h, and age-related macular degeneration: the Multi-ethnic Study of Atherosclerosis. Ophthalmology. 2008 Oct;115(10):1742-9. doi: 10.1016/j.ophtha.2008.03.021. Epub 2008 Jun 5. PMID 18538409
- [Result] Nguyen TT, Alibrahim E, Islam FM, Klein R, Klein BE, Cotch MF, Shea S, Wong TY. Inflammatory, hemostatic, and other novel biomarkers for diabetic retinopathy: the multi-ethnic study of atherosclerosis. Diabetes Care. 2009 Sep;32(9):1704-9. doi: 10.2337/dc09-0102. Epub 2009 Jun 23. PMID 19549733
- [Result] Kawasaki R, Cheung N, Islam FM, Klein R, Klein BE, Cotch MF, Sharrett AR, O'Leary D, Wong TY; Multi-Ethnic Study of Atherosclerosis. Is diabetic retinopathy related to subclinical cardiovascular disease? Ophthalmology. 2011 May;118(5):860-5. doi: 10.1016/j.ophtha.2010.08.040. Epub 2010 Dec 18. PMID 21168222
- [Result] Kreis AJ, Wong TY, Islam FM, Klein R, Klein BE, Cotch MF, Jenkins AJ, Shea S, Wang JJ. Is nuclear magnetic resonance lipoprotein subclass related to diabetic retinopathy? The multi-ethnic study of atherosclerosis (MESA). Diab Vasc Dis Res. 2009 Jan;6(1):40-2. doi: 10.3132/dvdr.2009.008. PMID 19156628
- [Result] Anuradha S, Healy GN, Dunstan DW, Klein R, Klein BE, Cotch MF, Wong TY, Owen N. Physical activity, television viewing time, and retinal microvascular caliber: the multi-ethnic study of atherosclerosis. Am J Epidemiol. 2011 Mar 1;173(5):518-25. doi: 10.1093/aje/kwq412. Epub 2011 Feb 7. PMID 21300854
- [Result] Greenstein MB, Myers CE, Meuer SM, Klein BE, Cotch MF, Wong TY, Klein R. Prevalence and characteristics of choroidal nevi: the multi-ethnic study of atherosclerosis. Ophthalmology. 2011 Dec;118(12):2468-73. doi: 10.1016/j.ophtha.2011.05.007. Epub 2011 Aug 4. PMID 21820181
- [Result] Ng CH, Cheung N, Wang JJ, Islam AF, Kawasaki R, Meuer SM, Cotch MF, Klein BE, Klein R, Wong TY. Prevalence and risk factors for epiretinal membranes in a multi-ethnic United States population. Ophthalmology. 2011 Apr;118(4):694-9. doi: 10.1016/j.ophtha.2010.08.009. Epub 2010 Oct 29. PMID 21035863
- [Result] Klein R, Klein BE, Knudtson MD, Wong TY, Cotch MF, Liu K, Burke G, Saad MF, Jacobs DR Jr. Prevalence of age-related macular degeneration in 4 racial/ethnic groups in the multi-ethnic study of atherosclerosis. Ophthalmology. 2006 Mar;113(3):373-80. doi: 10.1016/j.ophtha.2005.12.013. PMID 16513455
- [Result] Wong TY, Liew G, Tapp RJ, Schmidt MI, Wang JJ, Mitchell P, Klein R, Klein BE, Zimmet P, Shaw J. Relation between fasting glucose and retinopathy for diagnosis of diabetes: three population-based cross-sectional studies. Lancet. 2008 Mar 1;371(9614):736-43. doi: 10.1016/S0140-6736(08)60343-8. PMID 18313502
- [Result] Wong TY, Cheung N, Islam FM, Klein R, Criqui MH, Cotch MF, Carr JJ, Klein BE, Sharrett AR. Relation of retinopathy to coronary artery calcification: the multi-ethnic study of atherosclerosis. Am J Epidemiol. 2008 Jan 1;167(1):51-8. doi: 10.1093/aje/kwm256. Epub 2007 Sep 24. PMID 17893402
- [Result] Nguyen TT, Wang JJ, Sharrett AR, Islam FM, Klein R, Klein BE, Cotch MF, Wong TY. Relationship of retinal vascular caliber with diabetes and retinopathy: the Multi-Ethnic Study of Atherosclerosis (MESA). Diabetes Care. 2008 Mar;31(3):544-9. doi: 10.2337/dc07-1528. Epub 2007 Dec 10. PMID 18070990
- [Result] Cheung N, Bluemke DA, Klein R, Sharrett AR, Islam FM, Cotch MF, Klein BE, Criqui MH, Wong TY. Retinal arteriolar narrowing and left ventricular remodeling: the multi-ethnic study of atherosclerosis. J Am Coll Cardiol. 2007 Jul 3;50(1):48-55. doi: 10.1016/j.jacc.2007.03.029. Epub 2007 Jun 18. PMID 17601545
- [Result] Yau JW, Xie J, Lamoureux E, Klein R, Klein BE, Cotch MF, Bertoni AG, Shea S, Wong TY. Retinal microvascular calibre and risk of incident diabetes: the multi-ethnic study of atherosclerosis. Diabetes Res Clin Pract. 2012 Feb;95(2):265-74. doi: 10.1016/j.diabres.2011.10.027. Epub 2011 Nov 15. PMID 22088792
- [Result] Kawasaki R, Xie J, Cheung N, Lamoureux E, Klein R, Klein BE, Cotch MF, Sharrett AR, Shea S, Wong TY; MESA. Retinal microvascular signs and risk of stroke: the Multi-Ethnic Study of Atherosclerosis (MESA). Stroke. 2012 Dec;43(12):3245-51. doi: 10.1161/STROKEAHA.112.673335. Epub 2012 Oct 30. PMID 23111439
- [Result] Nguyen TT, Islam FM, Farouque HM, Klein R, Klein BE, Cotch MF, Herrington DM, Wong TY. Retinal vascular caliber and brachial flow-mediated dilation: the Multi-Ethnic Study of Atherosclerosis. Stroke. 2010 Jul;41(7):1343-8. doi: 10.1161/STROKEAHA.110.581017. Epub 2010 May 27. PMID 20508189
- [Result] Wong TY, Islam FM, Klein R, Klein BE, Cotch MF, Castro C, Sharrett AR, Shahar E. Retinal vascular caliber, cardiovascular risk factors, and inflammation: the multi-ethnic study of atherosclerosis (MESA). Invest Ophthalmol Vis Sci. 2006 Jun;47(6):2341-50. doi: 10.1167/iovs.05-1539. PMID 16723443
- [Result] Kawasaki R, Cheung N, Wang JJ, Klein R, Klein BE, Cotch MF, Sharrett AR, Shea S, Islam FA, Wong TY. Retinal vessel diameters and risk of hypertension: the Multiethnic Study of Atherosclerosis. J Hypertens. 2009 Dec;27(12):2386-93. doi: 10.1097/HJH.0b013e3283310f7e. PMID 19680136
- [Result] Ojaimi E, Nguyen TT, Klein R, Islam FM, Cotch MF, Klein BE, Wang JJ, Wong TY. Retinopathy signs in people without diabetes: the multi-ethnic study of atherosclerosis. Ophthalmology. 2011 Apr;118(4):656-62. doi: 10.1016/j.ophtha.2010.08.007. Epub 2010 Nov 4. PMID 21055817
- [Result] Klein R, Klein BE, Knudtson MD, Cotch MF, Wong TY, Liu K, Burke GL, Saad MF, Jacobs DR Jr, Sharrett AR. Subclinical atherosclerotic cardiovascular disease and early age-related macular degeneration in a multiracial cohort: the Multiethnic Study of Atherosclerosis. Arch Ophthalmol. 2007 Apr;125(4):534-43. doi: 10.1001/archopht.125.4.534. PMID 17420374
- [Result] Cheung N, Klein R, Wang JJ, Cotch MF, Islam AF, Klein BE, Cushman M, Wong TY. Traditional and novel cardiovascular risk factors for retinal vein occlusion: the multiethnic study of atherosclerosis. Invest Ophthalmol Vis Sci. 2008 Oct;49(10):4297-302. doi: 10.1167/iovs.08-1826. Epub 2008 Jun 6. PMID 18539932
- [Result] Fisher DE, Shrager S, Shea SJ, Burke GL, Klein R, Wong TY, Klein BE, Cotch MF. Visual Impairment in White, Chinese, Black, and Hispanic Participants from the Multi-Ethnic Study of Atherosclerosis Cohort. Ophthalmic Epidemiol. 2015;22(5):321-32. doi: 10.3109/09286586.2015.1066395. PMID 26395659